CLINICAL TRIAL: NCT01079689
Title: Brain Activity Changes Measured by EEG and fMRI on Healthy Volunteers After Complex Somatosensory Stimulation With Acupuncture Needles
Brief Title: Brain Activity Changes Measured by EEG and fMRI on Healthy Volunteers After Complex Somatosensory Stimulation
Acronym: BANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Max Planck Institute for Human Cognitive and Brain Sciences (Other); Berlin (Unknown)
Responsible Party: Principal Investigator, Claudia M. Witt, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: BANS10
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Healthy Volunteers
Keywords: basic science; healthy volunteers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: needle stimulation — stimulation with acupuncture needles

SUMMARY:
The purpose of this study is to evaluate effects on the brain after complex somatosensory stimulation with acupuncture needle. EEG and fMRI measurements will be performed.

DETAILED DESCRIPTION:
The aim of the study is to evaluate whether the point locations chosen for a complex somatosensory stimulation with acupuncture needles have an essential impact on the change of brain activity in healthy volunteers. For this, the investigators compare three different point locations (one acupuncture point and two non-acupuncture points) stimulated with acupuncture needles. Two measurements each with 20 subjects are planned.

* With the EEG measurements the impact of the stimulation's location on background rhythm especially in the somatosensoric cortex is evaluated.
* With the fMRI (functional magnetic resonance imaging) measurements the impact of the stimulation's location on BOLD (Blood Oxygen Level Dependency) signals and on functional connectivity is evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. healthy subjects of age from 18 to 40 years (inclusive)
2. right-handed (evaluated by "The Edinburgh Inventory")
3. with informed consent signed
4. no acupuncture treatment in the last 12 months
5. no medical knowledge about acupuncture
6. free time to take part in the measurements

Exclusion Criteria:

1. history of neurological and/or psychiatric diseases
2. history of brain injury
3. cognitive handicap, severe speech disorder, alcohol or drug abuse
4. history of neurosurgical intervention
5. chronic disease (e.g., asthma, diabetes mellitus etc.) with regular use of medications
6. pregnancy (tested by urine pregnancy test before the measurement) or planned pregnancy
7. any contraindication for acupuncture (e.g., anti-coagulation therapy)

   Additional exclusion criteria for fMRI measurement:
8. any contraindication for MRI (e.g., pacemaker, claustrophobia, cochlear implant, metallic implants etc. )

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Change in brain background rhythms after stimulation (baseline vs. post stimulation) in comparison between the three different point locations. | 26 minutes
Changes in resting state functional connectivity after stimulation (baseline vs. post-stimulation) in comparison between the three different point locations | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Max Planck Institute for Human Cognitive and Brain Sciences, Leipzig, Leipzig, Germany

REFERENCES:
- [Derived] Long X, Huang W, Napadow V, Liang F, Pleger B, Villringer A, Witt CM, Nierhaus T, Pach D. Sustained Effects of Acupuncture Stimulation Investigated with Centrality Mapping Analysis. Front Hum Neurosci. 2016 Oct 18;10:510. doi: 10.3389/fnhum.2016.00510. eCollection 2016. PMID 27803655